CLINICAL TRIAL: NCT07269184
Title: Impact of Ultrasound Guidance on Central Neuraxial Block Success in Patients With Non-Palpable Vertebral Anatomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, BURCUCAN, Asist. Doctor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2025-SEAH-BC-EA-palpation
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Epidural Analgesia; Ultrasound Assistance
Keywords: epidural; ultrasound; non-palpable spinous processes
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonography (U) (Active Comparator)
  Interventions: Procedure: epidural catheter, ultrasonography
- Palpation (P) (Active Comparator)
  Interventions: Procedure: anatomic landmark, epidural cateterisation

INTERVENTIONS:
Procedure: epidural catheter, ultrasonography — In the Ultrasound Group, surface marking will be performed in the operating room using ultrasonography.
  In the Anatomical Landmark Group, after the patient is positioned sitting in the operating room, the insertion site will be estimated by palpation of anatomical landmarks.
  Arms: Ultrasonography (U)
Procedure: anatomic landmark, epidural cateterisation — In the palpation group, after the patients are brought into the operating room and positioned sitting, the needle insertion site for epidural catheter placement will be determined by manual palpation
  Arms: Palpation (P)

SUMMARY:
Patients scheduled to undergo general surgery with planned epidural catheter placement will be evaluated by comparing two different techniques routinely used in anesthesia practice for catheter insertion.

A total of 60 patients aged 18-60 years, classified as ASA I-III, and scheduled to undergo general surgical procedures with epidural catheter placement at Sakarya University Faculty of Medicine Training and Research Hospital will be included in the study. All patients will be classified according to the following palpation scoring system to assess the difficulty of vertebral palpation:

Palpation Score: All patients will be evaluated in the sitting position, and the difficulty of palpating vertebral landmarks will be scored between 0 and 3:

0: Spinous processes and interspinous spaces are clearly identifiable

1. Spinous processes are palpable, but interspinous spaces are not clearly identifiable
2. Spinous processes are not palpable, interspinous spaces are not identifiable, but the vertebral column can be palpated either on or off the midline
3. Spinous processes and interspinous spaces are not palpable, and vertebral structures are not clearly distinguishable Patients with a palpation score of 3 will be included in the study group. Patients with a score of 0 will be included as the control group.

Patients will be divided into two groups: Anatomical Landmark Group and Ultrasound Group.

In the Ultrasound Group, surface marking will be performed in the operating room using ultrasonography.

In the Anatomical Landmark Group, after the patient is positioned sitting in the operating room, the insertion site will be estimated by palpation of anatomical landmarks.

After determining the needle entry point in both groups, epidural catheterization will be performed under sterile conditions according to our routine practice. The two groups will be compared in terms of first-attempt success rate, total procedure time, number of needle redirections, and complications occurring during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective general surgery
* Planned epidural catheterization
* Aged 18-60 years
* ASA physical status I-III
* Spinous processes not palpable (class3)

Exclusion Criteria:

* Contraindication to epidural catheterization
* ASA physical status IV-V
* Diagnosed with scoliosis
* Presence of anatomical deformities
* Declining to participate in the study
* Patients for whom follow-up conditions cannot be ensured

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
first-attempt success rate | 3 months